CLINICAL TRIAL: NCT01845714
Title: Impact of Keratoconus, Cross-linking and Cross-linking Combined With Topo-guided Photorefractive Keratectomy on Self-reported Quality of Life. A Three-year Update.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Assistant Professor, Democritus University of Thrace
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EIT-KC-VSQOL3
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Keratoconus
Keywords: Keratoconus; Corneal cross Linking; Topo guided PRK; Quality of Life
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Cross Linking Group (CxL group) (Active Comparator): Patients that received CXL
  Interventions: Procedure: Corneal Cross Linking
- Cross Linking with topo-guided PRK (tCxL) (Active Comparator): Patients that received tCxL
  Interventions: Procedure: Corneal Cross Linking combined with topoguided PRK

INTERVENTIONS:
Procedure: Corneal Cross Linking
  Arms: Cross Linking Group (CxL group)
Procedure: Corneal Cross Linking combined with topoguided PRK
  Arms: Cross Linking with topo-guided PRK (tCxL)

SUMMARY:
Study Hypothesis: Former investigators indicated that keratoconus has a negative impact on vision-specific quality of life. This study attempts to confirm this statement and assess whether cross-linking and cross-linking combined with photorefractive keratectomy improve vision-specific quality of life, in a sample of keratoconus patients with 3-years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* be diagnosed and classified as stage 1 keratoconus according to the Amsler-Krumeich classification system for keratoconus
* present progressive keratoconus in consecutive corneal topographies, and/or changes in their refractive power.

Progressive keratoconus was defined when any of the following criteria was met for a period of 24 months:

* an increase of 1.00 diopter (D) or more in the steepest keratometry measurement
* an increase of 1.00 D or more in manifest cylinder
* an increase of 0.50 D or more in manifest refraction spherical equivalent.

Exclusion Criteria:

* glaucoma
* suspicion for glaucoma
* IOP-lowering medications
* central corneal thickness (CCT) less than 400μm
* K-readings more than 60D
* history of herpetic keratitis
* corneal scarring
* severe eye dryness
* pregnancy or nursing
* current corneal infection
* or underlying autoimmune disease KG members were further sub-divided into CxL and tCxL groups, according to their eligibility for treatment with CxL or CxL with tPRK. In order to be eligible for tCxL, group participants should, additionally, have CCT above 450μm.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Vision Specific quality of Life (VS-QoL) | 3 years

REFERENCES:
- [Result] Labiris G, Giarmoukakis A, Sideroudi H, Kozobolis V. Impact of keratoconus, cross-linking and cross-linking combined with topography-guided photorefractive keratectomy on self-reported quality of life: a 3-year update. Cornea. 2013 Sep;32(9):e186-8. doi: 10.1097/ICO.0b013e318296e13c. No abstract available. PMID 23807006